CLINICAL TRIAL: NCT00866437
Title: Prospective, Controlled, Single-blinded, Longitudinal, Two-arms, Clinical Study Evaluation of Efficacy/Safety of EVE-PMS Skin-Test Panel -Detecting Sensitivity to Sex Hormones in Women With Premenstrual Syndrome
Brief Title: Evaluation of Efficacy/Safety of EVE-PMS Skin Test Panel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EVE Medical Systems Ltd. (Industry)
Responsible Party: Dr. Yonit Bomstein, EVE Medical Systems Ltd.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: EveMS-0908
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-02

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; Hormones; Skin tests; Allergen Immunotherapy
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Progesterone; Estradiol; Estrone; Estriol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Control group (Experimental)
  Interventions: Drug: Skin test panel
- PMS (Experimental)
  Interventions: Drug: Skin test panel

INTERVENTIONS:
Drug: Skin test panel — Skin testing 4 sex hormones will be performed during the luteal phase of the subject's menstrual cycle by study investigators.
  Hormones:
  1. Progesterone 1mmol/L
  2. Estradiol 1mmol/L
  3. Estrone 3mmol/L
  4. Estriol 3mmol/l
     Controls:
  5. Saline (NaCl) 0.9%
  6. Ethyl Oleate with 10% Benzyl Alcohol
  7. Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Other Names: Progesterone; Estradiol; Estrone; Estriol
  Arms: Healthy Control group
Drug: Skin test panel — Hormones:
  1. Progesterone 1mmol/L
  2. Estradiol 1 mmol/L
  3. Estrone 3 mmol/L
  4. Estriol 3mmol/l
     Controls:
  5. Saline (NaCl) 0.9%
  6. Ethyl Oleate with 10% Benzyl Alcohol
  7. Histamine phosphate 1mg/ml (epicutaneous- prick test)
  Other Names: Progesterone; Estradiol; Estrone; Estriol
  Arms: PMS

SUMMARY:
The EVE-PMS technology is intended for determination of intolerance or sensitivity to sex hormones, among women suffering from severe PreMenstrual Syndrome (PMS).

The system includes skin testing panel for identification of hormones to which the patients might be sensitive. Tests are applied close to the ovulation period and the skin reaction is examined in 20 minutes, 48 hours and daily during the following month. Results of skin tests and patient's history will determine the value of EVE-PMS Skin-Test Panel as a diagnostic tool for severe PMS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Person is over the age of 20 but not older than age 45.
2. Person is willing to participate as evidenced by signing the written informed consent form.
3. Suffers from known dominant severe symptom of breast swelling and tenderness (level 7-10 according to standard scale of PMS symptoms severity)
4. Other severe symptoms of Premenstrual syndrome (based on WHO and ACOG criteria). This may include one or more of PMS symptoms with level 7-10 according to standard scale of PMS symptoms severity.
5. At work, school, home, or in daily routine, at least one of the PMS symptoms caused reduction of productivity or inefficiency
6. At least one of the PMS symptoms caused avoidance of or less participation in hobbies or social activities
7. At least one of the PMS symptoms interfere with relationships with others:

   i. Timing of PMS symptom(s): during the 14 days prior to onset of menstrual flow (rather than spotting) and up to 5 days during the menstrual flow.

ii. Pattern and length of PMS symptomatic period: minimum of 2 days, up to 14 days.

iii. For PMS diagnosis two out of last three consecutive menstrual cycles were monitored by daily monitoring of symptoms.

iv. Timing and length of asymptomatic phase: day 6 to at least day 10 of the menstrual cycle.

v. Cyclicity - presentation of the 'off-on' phenomenon: there should be a clear shift from no PMS symptoms to PMS symptoms.

vi. Reliable non hormonal contraception.

Exclusion Criteria:

1. Pregnant or lactating woman
2. Oral contraceptives during last three months, including hormonal IUD (trade name mirena).
3. Serious health problems.
4. Unexplained menstrual disorders.
5. Treated by hormones (estrogen and progesterone).
6. For healthy: Irregular or abnormal test results.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
EVE-PMS Skin-Test Panel can obtain statistically significant sensitivity & specificity to support the diagnosis of PMS, particularly in women with severe symptoms(i.e. breast swelling; tenderness; other PMS symptoms according to widely accepted criteria | Total study duration will be approximately 2-3 months

SECONDARY OUTCOMES:
Minimal skin test related adverse events. | 2-3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Avner Reshef, Dr., Principal Investigator — Allergy and clinical Immunology Department
Locations (1):
- Sheba Medical Center, Tel-Hashomer, Ramat Efal, Israel